CLINICAL TRIAL: NCT01795495
Title: Analgesia Following Posterior Spinal Fusion: Methadone vs Magnesium
Brief Title: Methadone vs Magnesium in Spinal Fusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, David P. Martin, Clinical Assistant Professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB13-0036; Active (Other Grant/Funding Number: Nationwide Children's Hospital Intramural Grant - 292913)
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Idiopathic Scoliosis
Keywords: Spinal Fusion; Scoliosis; Methadone; Magnesium; Adolescents; Back Surgery
MeSH Terms: conditions — Scoliosis | interventions — Methadone; Magnesium Sulfate; Magnesium; Remifentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Remifentanil (Active Comparator): This arm will receive remifentanil alone as is the current practice.
  Interventions: Drug: Remifentanil
- Remifentanil plus methadone (Experimental): This arm will receive the current analgesic remifentanil plus and adjunct dose of methadone hydrochloride.
  Interventions: Drug: Methadone hydrochloride
- Remifentanil plus magnesium (Experimental): This arm will receive the current analgesic remifentanil plus an adjunct dose of magnesium sulfate.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Methadone hydrochloride — This drug will be used in conjunction with remifentanil as an adjunct analgesic. Remifentanil + methadone (0.1 mg/kg IV over 15 minutes) just after induction of anesthesia
  Other Names: Methadone
  Arms: Remifentanil plus methadone
Drug: Magnesium Sulfate — This drug will be given with remifentanil as an adjunct analgesic. Remifentanil + magnesium (50 mg/kg bolus over 30 minutes followed by 10 mg/kg/hour).
  Other Names: Magnesium
  Arms: Remifentanil plus magnesium
Drug: Remifentanil
  Arms: Remifentanil

SUMMARY:
Significant pain may occur following posterior spinal fusion despite the use of conventionally accepted techniques including patient controlled analgesia. If detected, a significant reduction in opioid requirements may lead to improved patient satisfaction and decreased opiate side effects.

The current study would use a prospective, randomized trial investigating the efficacy of one of 2 regimens as adjuncts to intraoperative anesthesia and postoperative analgesia, along with a third control group. The patients would be randomized to receive remifentanil plus a single intraoperative dose of methadone; remifentanil plus a bolus followed by an infusion of magnesium; or remifentanil alone. In addition, the two medications being studied might make it easier to determine the efficacy of neurophysiologic monitoring including somatosensory evoked potential (SSEP) (amplitude and latency) and motor evoked potential (MEP) (mA) required to elicit the response.

The purpose of this study would be to explore the effects of intraoperative methadone vs magnesium on intraoperative anesthetic requirements, postoperative opioid requirements, the efficacy of neurophysiologic monitoring including SSEP and MEP, inspired concentration of desflurane, remifentanil, and the need for intraoperative supplemental agents to control blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 12, and younger than 19 years of age undergoing posterior spinal fusion for idiopathic scoliosis
* American Society of Anesthesiologist (ASA) physical status I or II
* Parents/Guardian willing and able to authorize informed consent
* Patients willing and able to authorize assent

Exclusion Criteria:

* Patients presenting with neuromuscular scoliosis
* Patients deemed at increased risk of adverse reactions due to the presence of pre-existing severe organ system dysfunction, including debilitating lung disease, severe obstructive sleep apnea, severe congenital or acquired heart disease, and/or severe renal impairment
* Patients who are both being currently treated for a psychological disorder and have a history of hospitalization for said disorder

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2013-09; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P. Martin, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Stemland CJ, Witte J, Colquhoun DA, Durieux ME, Langman LJ, Balireddy R, Thammishetti S, Abel MF, Anderson BJ. The pharmacokinetics of methadone in adolescents undergoing posterior spinal fusion. Paediatr Anaesth. 2013 Jan;23(1):51-7. doi: 10.1111/pan.12021. Epub 2012 Sep 14. PMID 22978825
- [Background] Sharma A, Tallchief D, Blood J, Kim T, London A, Kharasch ED. Perioperative pharmacokinetics of methadone in adolescents. Anesthesiology. 2011 Dec;115(6):1153-61. doi: 10.1097/ALN.0b013e318238fec5. PMID 22037641
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Elsharnouby NM, Elsharnouby MM. Magnesium sulphate as a technique of hypotensive anaesthesia. Br J Anaesth. 2006 Jun;96(6):727-31. doi: 10.1093/bja/ael085. Epub 2006 May 2. PMID 16670112
- [Background] Levaux Ch, Bonhomme V, Dewandre PY, Brichant JF, Hans P. Effect of intra-operative magnesium sulphate on pain relief and patient comfort after major lumbar orthopaedic surgery. Anaesthesia. 2003 Feb;58(2):131-5. doi: 10.1046/j.1365-2044.2003.02999.x. PMID 12562408
- [Derived] Martin DP, Samora WP 3rd, Beebe AC, Klamar J, Gill L, Bhalla T, Veneziano G, Thung A, Tumin D, Barry N, Rice J, Tobias JD. Analgesic effects of methadone and magnesium following posterior spinal fusion for idiopathic scoliosis in adolescents: a randomized controlled trial. J Anesth. 2018 Oct;32(5):702-708. doi: 10.1007/s00540-018-2541-5. Epub 2018 Aug 4. PMID 30078167

RESULTS

PARTICIPANT FLOW:
Groups:
- Remifentanil: This arm will receive remifentanil alone as is the current practice.
  Remifentanil
Period: Overall Study
Arm/Group | Remifentanil | Remifentanil Plus Methadone | Remifentanil Plus Magnesium
Started | 20 | 22 | 21
Completed | 19 | 22 | 19
Not Completed | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil | Remifentanil Plus Methadone | Remifentanil Plus Magnesium | Total
Number analyzed (Participants) | 20 | 22 | 21 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (1.4) | 15.4 (1.2) | 15.3 (1.9) | 15.0 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 18 | 52
  Male | 3 | 5 | 3 | 11
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 21.6 (4.3) | 22.8 (5.7) | 24.2 (5.6) | 22.6 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Intra- and Post-operative Pain Relief
Description: To prospectively compare the effects of intra-operative methadone and magnesium on postoperative opioid requirements. Total amount of hydromorphone administered in OR, recovery room (PACU), and on the inpatient ward 24 hours post-operatively.
Time Frame: Intra-operative and 24 hours post-operatively
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Remifentanil | Remifentanil Plus Methadone | Remifentanil Plus Magnesium
Number analyzed (Participants) | 19 | 22 | 19
mg/kg | 0.34 (0.11) | 0.26 (0.1) | 0.38 (0.1)

2. Secondary Outcome: Post-operative Pain Scores
Description: VAS pain score - 0 being no pain and 10 being worst pain.
Time Frame: Post-operatively to 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remifentanil | Remifentanil Plus Methadone | Remifentanil Plus Magnesium
Number analyzed (Participants) | 19 | 22 | 19
units on a scale | 4.6 (2.2) | 5.1 (1.8) | 5.1 (1.2)

ADVERSE EVENTS:
Arm/Group | Remifentanil | Remifentanil Plus Methadone | Remifentanil Plus Magnesium
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes